CLINICAL TRIAL: NCT03869775
Title: Observational Study Relationship Between Perfusion Index Changes and Intraoperative Complications in Cardiovascular Autonom Neuropathia Type-2 DM Patients With Spinal Anesthesia
Brief Title: Perfusion Index Changes in Cardiovascular Autonom Neuropathia Type-2 Dm Whit Spinal Anesthesia
Acronym: PI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, faruk subasi, Asistant Doctor, Erzincan University
Other Study IDs: ErzincanU
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia; Adverse Effect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- control group: no additional disease
  Interventions: Device: perfusion index monitor
- working group-1: additional disease only DM and no cardıovascular autonomous neuropathıa
  Interventions: Device: perfusion index monitor; Diagnostic Test: ewing test
- working group-2: additional disease only DM and pozitif cardıovascular autonomous neuropathıa
  Interventions: Device: perfusion index monitor; Diagnostic Test: ewing test

INTERVENTIONS:
Device: perfusion index monitor — perfusion index measured in patients undergoing spinal anesthesia with non-invasive perfusion index monitor
Diagnostic Test: ewing test — ewing tests will be applied to diabetic patients undergoing spinal anesthesia for cardıovascular autonomous neuropathıa diagnosis
  Groups: working group-1; working group-2

SUMMARY:
Cardiovascular autonomic neuropathy in diabetic patients, hypertension, sympathovagal imbalance, orthostatic hypotension, painless myocardial infarction, ischemia, left ventricular dysfunction, cardiac sympathetic and parasympathetic innervation disturbances, qt interval prolongation and sudden deaths observed. The purpose of this study is to evaluate the relationship between cardiovascular autonomic neuropathy and perfusion index in spinal anesthesia

DETAILED DESCRIPTION:
Cardiovascular autonomic neuropathy in diabetic patients, hypertension, sympathovagal imbalance, orthostatic hypotension, painless myocardial infarction, ischemia, left ventricular dysfunction, cardiac sympathetic and parasympathetic innervation disturbances, qt interval prolongation and sudden deaths observed. The purpose of this study is to evaluate the relationship between cardiovascular autonomic neuropathy and perfusion index in spinal anesthesia

ELIGIBILITY:
Inclusion Criteria:

* the patient will be operated with spinal anesthesia
* over 18 years
* no additional disease and only DM

Exclusion Criteria:

* patients with additional disease
* patients under 18 years of age
* patients contraindicated in spinal anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years old
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Perfusion index change | Day 1
  Perfusion index change in spinal anesthesia related cardiovascular autonom neuropatia

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincanu, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided